CLINICAL TRIAL: NCT02893254
Title: A Multicenter, Randomized, Double-blind, Parallel-controlled Phase 3 Study Evaluating the Efficacy and Safety of Recombinant Human Monoclonal Antibody Against Human Tumor Necrosis Factor-α (IBI303) Compared to Adalimumab in Patients With Active Ankylosing Spondylitis
Brief Title: Efficacy and Safety of IBI303 in Adult Patients With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI303A301
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: AS
Keywords: ankylosing spondylitis, tumor necrosis factor-α inhibitors
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IBI303 (Experimental): IBI303 40mg administered subcutaneously every other week, 12cycles
  Interventions: Drug: IBI303
- Adalimumab (Active Comparator): Adalimumab 40mg administered subcutaneously every other week
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: IBI303 — 12 cycles. IBI303: 40 mg, iH
  Arms: IBI303
Drug: Adalimumab — 12 cycles. Adalimumab: 40mg, iH
  Arms: Adalimumab

SUMMARY:
Study of the efficacy and safety of IBI303 compared with adalimumab in adult patients with ankylosing spondylitis (AS) who have had an inadequate response to or who are intolerant to one or more nonsteroidal anti-inflammatory drugs (NSAIDs)

DETAILED DESCRIPTION:
Adults patients with active ankylosing spondylitis (AS) were randomized in a 1:1 ratio to receive treatment with adalimumab 40 mg every other week (eow) or IBI303, given subcutaneously (SC), in the 24-week double-blind (DB) phase. Randomized participants received one SC injection of the appropriate DB study medication (adalimumab 40 mg or IBI303) at Week 0 and then eow until Week 22. A follow-up visit occurred 70 days(Week 32) after the last dose of study drug to obtain information on any ongoing or new adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 65 years of age
2. Fulfilled modified New York Criteria for AS, had active disease（as defined by≥2 of the following: Bath AS Disease Activity Index(BASDAI) ≥4(10cm VAS); total back pain≥40(100mm VAS) and ≥1 hour of morning stiffness）
3. No response, or inadequate response, or intolerant to≥1 NSAID at least 4 weeks
4. Participants who are regularly taking DMARDs(SSZ≤3g/day，MTX≤15mg/week) as part of their AS therapy are required to be on a stable dose ≥28 days prior to Baseline, and are required to be on a stable DMARDs dose and to accept oral folic acid therapy(≥5mg/week) during the study period；
5. Participants who are regularly taking NSAIDs as part of their AS therapy are required to be on a stable dose ≥14 days prior to Baseline, and are required to be on a stable dose during the study period；
6. Glucocorticoid must be withdrawn for at least 4 weeks prior to Baseline, and were not allowed during the study period.
7. Total duration of prior physical therapy should be at least 2 weeks
8. Traditional Chinese medicines to AS must be withdrawn for at least 28 days prior to Baseline, and were not allowed during the study period.
9. Biological agents must be withdrawn: etanercept and anakinra(IL-1 receptor antagonist) for at least 4 weeks prior to administration; tocilizumab(IL-6 monoclonal antibody) for at least 12 weeks prior to administration; other biological agents for 12 weeks or 5 half-lives(whichever is longer) prior to administration
10. Male subjects' partner, or female subjects should be willing to use adequate contraception from admission to clinical research center until 5 months post dosing；
11. To fully understanding the purpose of the study, to understand the pharmacological action of the study drugs and the possible adverse reactions; participants who are voluntary to sign the informed consent according to the Declaration of Helsinki
12. Blood routine examination: hemoglobin ≥90g/L, WBC count ≥3.5×109/L, PLT count ≥100×109/L; liver function examination: total bilirubin(TBIL), direct bilirubin(DBIL), aspartate transaminase(AST) or alanine aminotransferase (ALT) <1.5×ULN; kidney function examination：creatinine(Cr) ≤ULM, usea nitrogen(BUN) ≤1.25×ULN

Exclusion Criteria:

1. No response to prior tumor necrosis factor-α inhibitors treatment
2. Use of DMARD(except for sulfasalazine or methotrexate) within 4 weeks prior to Baseline
3. Use of opioid analgesics(such as methadone, morphine) within 4 weeks prior to Baseline
4. X-ray suggests total spinal ankylosis, or sacroiliac joint fusion
5. Patients with moderate to severe congestive heart failure（NYHA ）
6. Has received intra-articular joint injection(s), spinal or paraspinal injection(s) with corticosteroids within 28 days prior to Baseline
7. Has undergone spinal surgery or joint surgery within 2 months prior to the administration of the study drugs
8. Patients with other rheumatic diseases or immunodeficiency, including inflammatory bowel disease(IBD), psoriasis, active uveitis
9. Recent active or chronic infection requiring anti-infective therapy, such as M.tuberculosis, Listeriosis, Histophasmosis
10. Tuberculosis(TB) history, or a positive T-SPOT test, or chest radiograph suggests active TB
11. Positive serology for human immunodeficiency virus(HIV) antibody
12. Positive serology for hepatitis C virus antibody
13. Active or chronic HBV infection, such as positive hepatitis B virus surface antigen
14. Malignancy history ≤5 years（except for successfully treated cutaneous squamous cell carcinoma, or basal cell carcinoma, or localized cervical carcinoma in situ, or breast ductal carcinoma in situ）
15. History of relevant allergy/hypersensitivity (including allergy to the study medications or its excipients)
16. Prior or recent central nervous system demyelinating disease or multiple sclerosis
17. Use of live vaccines within 3 months prior to Baseline
18. Pregnant or breastfeeding women
19. Suspected or confirmed drug/alcohol use
20. Participation in another interventional trial within 3 months prior to administration
21. Subjects with serious psychiatric or nervous system diseases, or patients who have difficulty in informing consent or AE presentation, or illiterate patients
22. Subjects who are unable to complete the study, or who may not be able to comply with the requirement of the study, judged by the investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Number of participants meeting the Assessment of Spondyloarthritis International Society(ASAS) ASAS20 Response Criteria | Week 24

SECONDARY OUTCOMES:
Number of participants meeting the ASAS20 Response | Week 2
Number of participants meeting the ASAS20 Response | Week 4
Number of participants meeting the ASAS20 Response | Week 8
Number of participants meeting the ASAS20 Response | Week 12
Number of participants meeting the ASAS20 Response | Week 16
Number of participants meeting the ASAS20 Response | Week 20
Number of participants meeting the ASAS40 Response Criteria | Week 24
Number of Participants Meeting the ASAS5/6 Response Criteria | Week 24
Number of Participants Meeting the ASAS Partial Remission | Week 24
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index(BASDAI), in Bath Ankylosing Spondylitis Functional Index(BASFI), in Bath Ankylosing Spondylitis Measure Index(BASMI) | Baseline and Week 24
Number of participants meeting the ASAS40 Response Criteria | Week 2
Number of participants meeting the ASAS40 Response Criteria | Week 4
Number of participants meeting the ASAS40 Response Criteria | Week 8
Number of participants meeting the ASAS40 Response Criteria | Week12
Number of participants meeting the ASAS40 Response Criteria | Week16
Number of participants meeting the ASAS40 Response Criteria | Week20
Number of Participants Meeting the ASAS5/6 Response Criteria | Week 2
Number of Participants Meeting the ASAS5/6 Response Criteria | Week 4
Number of Participants Meeting the ASAS5/6 Response Criteria | Week 8
Number of Participants Meeting the ASAS5/6 Response Criteria | Week 12
Number of Participants Meeting the ASAS5/6 Response Criteria | Week 16
Number of Participants Meeting the ASAS5/6 Response Criteria | Week 20
Number of Participants Meeting the ASAS Partial Remission | Week 2
Number of Participants Meeting the ASAS Partial Remission | Week 4
Number of Participants Meeting the ASAS Partial Remission | Week 8
Number of Participants Meeting the ASAS Partial Remission | Week 12
Number of Participants Meeting the ASAS Partial Remission | Week 16
Number of Participants Meeting the ASAS Partial Remission | Week 20
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index(BASDAI), in Bath Ankylosing Spondylitis Functional Index(BASFI), in Bath Ankylosing Spondylitis Messure Index(BASMI) | Baseline and Week 2
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index(BASDAI), in Bath Ankylosing Spondylitis Functional Index(BASFI), in Bath Ankylosing Spondylitis Messure Index(BASMI) | Baseline and Week 4
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index(BASDAI), in Bath Ankylosing Spondylitis Functional Index(BASFI), in Bath Ankylosing Spondylitis Messure Index(BASMI) | Baseline and Week 8
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index(BASDAI), in Bath Ankylosing Spondylitis Functional Index(BASFI), in Bath Ankylosing Spondylitis Messure Index(BASMI) | Baseline and Week 12
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index(BASDAI), in Bath Ankylosing Spondylitis Functional Index(BASFI), in Bath Ankylosing Spondylitis Messure Index(BASMI) | Baseline and Week 16
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index(BASDAI), in Bath Ankylosing Spondylitis Functional Index(BASFI), in Bath Ankylosing Spondylitis Messure Index(BASMI) | Baseline and Week 20
Change from Baseline in Patient Global Assessment of Disease Activity | Baseline and Week 12
Change from Baseline in Patient Global Assessment of Disease Activity | Baseline and Week 24
Change from Baseline in Total Back Pain Score | Baseline and Week 12
Change from Baseline in Total Back Pain Score | Baseline and Week 24
Change From Baseline in Inflammation Score | Baseline and Week 12
Change From Baseline in Inflammation Score | Baseline and Week 24
Change from Baseline in Maastricht Ankylosing Spondylitis Enthesis Score(MASES) | Baseline and Week 12
Change from Baseline in Maastricht Ankylosing Spondylitis Enthesis Score(MASES) | Baseline and Week 24
Change from Baseline in ASDAS-CRP and ASDAS-ESR | Baseline and Week 12
Change from Baseline in ASDAS-CRP and ASDAS-ESR | Baseline and Week 24
Change from Baseline in EQ-5D/WPAI-SHP/HAQ-S QoL | Baseline and Week 12
Change from Baseline in EQ-5D/WPAI-SHP/HAQ-S QoL | Baseline and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Huji Xu, Principal Investigator — Shanghai Changzheng Hospital

REFERENCES:
- [Result] Huang F, Gu J, Zhu P, Bao C, Xu J, Xu H, Wu H, Wang G, Shi Q, Andhivarothai N, Anderson J, Pangan AL. Efficacy and safety of adalimumab in Chinese adults with active ankylosing spondylitis: results of a randomised, controlled trial. Ann Rheum Dis. 2014 Mar;73(3):587-94. doi: 10.1136/annrheumdis-2012-202533. Epub 2013 Mar 8. PMID 23475983
- [Derived] Xu H, Li Z, Wu J, Xing Q, Shi G, Li J, Liu X, Wu L, Li X, Tan W, He D, Bi L, Li H, Xiao Z, Shuai Z, Li X, Wang Y, Luo L, Zheng Y, Xiao W, Wu X, Zhou L, Li T, Qian L, Zhou H, Lu S, Zheng S, Xiong Y, Wang X, Wang Y, Wu X. IBI303, a biosimilar to adalimumab, for the treatment of patients with ankylosing spondylitis in China: a randomised, double-blind, phase 3 equivalence trial. Lancet Rheumatol. 2019 Sep;1(1):e35-e43. doi: 10.1016/S2665-9913(19)30013-X. Epub 2019 Aug 28. PMID 38229357